CLINICAL TRIAL: NCT00997178
Title: A Multicenter Randomized Single-Masked Clinical Trial Testing the Effect of Non-surgical Periodontal Therapy on Glycosylated Hemoglobin (HbA1c) Levels in Subjects With Type 2 Diabetes and Chronic Periodontitis
Brief Title: Diabetes and Periodontal Therapy Trial
Acronym: DPTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Minnesota (Other); The University of Texas Health Science Center, Houston (Other); The University of Texas Health Science Center at San Antonio (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCR:07-003; U01DE018902-01 (NIH); U01DE018886-01 (NIH)
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes
Keywords: Diabetes; Diabetes Mellitus; Periodontal Disease; Periodontitis; Glycosylated Hemoglobin; HbA1c
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-surgical periodontal therapy (Experimental): Non-surgical periodontal therapy consisted of scaling and root planing plus chlorhexidine oral rinse at baseline and supportive periodontal therapy at 3 and 6 months
  Interventions: Procedure: Non-surgical periodontal therapy
- Delayed non-surgical periodontal therapy (Other): No periodontal treatment for 6 months
  Interventions: Other: Delayed non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — Non-surgical periodontal therapy (scaling and root planing)and supportive periodontal therapy with chlorhexidine rinse
  Arms: Non-surgical periodontal therapy
Other: Delayed non-surgical periodontal therapy — Delayed non-surgical periodontal therapy (scaling and root planing) after the 6 month visit
  Arms: Delayed non-surgical periodontal therapy

SUMMARY:
The primary aim of the study is to determine if non-surgical periodontal therapy (scaling and root planing and supportive periodontal therapy) is efficacious compared to delayed therapy in reducing elevated glycosylated hemoglobin (HbA1c) at 6 months post-randomization in subjects with type 2 diabetes and untreated, moderate to advanced chronic periodontitis.

The secondary aims of the study are to:

1. evaluate whether 6 month (or shorter-term (3 month)) changes in clinical measures of chronic periodontitis (gingival index, bleeding on probing, probing depth, clinical attachment level) are related to changes in HbA1c and fasting glucose or insulin resistance as measured by the Homeostasis Model Assessment 2 (HOMA2).
2. assess the 3 month and 6 month efficacy of periodontal therapy on all of the above study outcomes. If a treatment response is observed for any of the study outcomes at 3 months, then the trial can evaluate whether this response is sustained at 6 months.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled, single-masked, Phase III trial to determine if non-surgical periodontal therapy (scaling and root planing) is efficacious in reducing elevated glycosylated hemoglobin (HbA1c) at 6 months post-randomization in subjects with type 2 diabetes and untreated, moderate to advanced chronic periodontitis. Six hundred adults with a diagnosis of type 2 diabetes and chronic periodontitis will be randomized at three Clinical Sites; University of Alabama at Birmingham; the University of Minnesota, Minneapolis; and the University of Texas Health Science Center, San Antonio. The Core Laboratory will be located at the University of Minnesota and the Study Chair's Office and Coordinating Center will be located at Stony Brook University, Stony Brook, New York.

Eligible participants will be randomly assigned to receive either initial non-surgical periodontal therapy with chlorhexidine rinse (treatment subjects) or delayed non-surgical periodontal therapy (control subjects). Control subjects will be offered delayed periodontal therapy (scaling and root planing) following the 6 month visit. Participants meeting all other eligibility criteria and needing essential dental care, i.e., for broken, grossly carious or abscessed teeth, may enroll only following completion of necessary dental treatment. Participants in both study arms will receive oral hygiene instruction and healthy lifestyle information (e.g. diet, exercise) at baseline and at the 3 and 6 month visits.

Periodontal data will be recorded by trained and calibrated examiners at baseline and 3 and 6 months following randomization. Fasting blood will collected at baseline and at 3 and 6 months to measure intermediate links in the putative causal chain between periodontitis and glycemic control. The periodontal health of all subjects will be monitored, and any subject who experiences progressive periodontitis during the study will be provided with non-surgical rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years of age
* Screening HbA1c value ≥ 7% and <9%
* Physician diagnosed type 2 diabetes of more than three months duration
* Currently under the care of a physician for diabetes management
* No change in diabetes-related medications during the three months prior to enrollment. Change is defined as any of the following: change in dose of any 1 hyperglycemic drug by more than two-fold, change in dose of insulin of more than 10%, addition or subtraction of an oral hyperglycemic agent or insulin.
* Consent to contact treating physician and obtain physician agreement to refrain from changing diabetes- related medications during DPTT participation unless overt symptoms develop (e.g. polydipsia, polyuria), HbA1c is 9.5% or higher
* Moderate to severe chronic periodontitis, defined as loss of clinical attachment and probing depth of ≥5 mm at two sites in the mouth in 2 or more quadrants
* No definitive periodontal treatment during the six months prior to enrollment
* Likely to have at least 16 natural teeth for the entire length of study
* Informed consent obtained and signed
* Ability and willingness to cooperate with the study protocol and attend all study visits over the next 9 months
* Willingness to avoid pregnancy during study participation

Exclusion Criteria:

* Self-reported serious concurrent disease that at the discretion of the referring physician limits life expectancy to less than 1 year.
* Emergency room visit or physician visit within the last 30 days because of hyperglycemia or diabetes complications.
* Chronic or continuous use (daily for more than 7 consecutive days) of nonsteroidal anti-inflammatory drugs within the preceding 2 months, other than low dose aspirin (e.g. 75-325 mg/day).
* Receiving chronic treatment with systemic corticosteroids, cyclosporine or other systemic immunosuppressive drugs
* Chronic treatment with systemic antibiotics (antibiotics for > 7 consecutive days within 30 days of baseline visit).
* Currently receiving dialysis.
* At increased risk of bleeding complications from dental treatment, based on medical history.
* Requires Essential Dental Care (e.g., treatment for grossly decayed teeth, broken teeth, dental abscesses, peri-apical infections, other dental infections).
* Heavy alcohol consumption (on average > 2 drinks/day for women and > 3 drinks/day for men).
* Currently pregnant or considering becoming pregnant within the 6 month follow-up period
* Any other criteria that in the opinion of the investigator would preclude study completion or problems with compliance

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Hemoglobin (HbA1c) | 6 months after randomization

SECONDARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) | 3 months after randomization
Change in Fasting Plasma Glucose and Homeostasis Model Assessment 2 (HOMA2) | 3 and 6 months after randomization
Change in clinical measures of chronic periodontitis (gingival index, bleeding on probing, probing depth, clinical attachment level) | 3 and 6 months after randomization
Need for Periodontal Rescue Therapy | When required
Change in diabetes medications | 3 and 6 months after randomization
Need for Diabetes Rescue Therapy | When required

CONTACTS AND LOCATIONS:
Overall Officials: Steven Engebretson, DMD, MS, MS, Study Chair — Stony Brook University; Leslie Hyman, PhD, Study Director — Stony Brook University
Locations (8):
- United States (8):
  - Clinical Site: University of Alabama at Birmingham, Birmingham, Alabama
  - Clinical Site: University of Minnesota, Minneapolis, Minnesota
  - Core Laboratory: University of Minnesota, Minneapolis, Minnesota
  - Coordinating Center: Stony Brook University-, Stony Brook, New York
  - Administrative Center/Study Chair's Office: Stony Brook University, Stony Brook, New York
  - Clinical Site: Stony Brook University, Stony Brook, New York
  - University of Texas, Health Sciences Center at Houston, Houston, Texas
  - Clinical Site: University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Result] Engebretson SP, Hyman LG, Michalowicz BS, Schoenfeld ER, Gelato MC, Hou W, Seaquist ER, Reddy MS, Lewis CE, Oates TW, Tripathy D, Katancik JA, Orlander PR, Paquette DW, Hanson NQ, Tsai MY. The effect of nonsurgical periodontal therapy on hemoglobin A1c levels in persons with type 2 diabetes and chronic periodontitis: a randomized clinical trial. JAMA. 2013 Dec 18;310(23):2523-32. doi: 10.1001/jama.2013.282431. PMID 24346989
- [Derived] Geisinger ML, Michalowicz BS, Hou W, Schoenfeld E, Gelato M, Engebretson SP, Reddy MS, Hyman L. Systemic Inflammatory Biomarkers and Their Association With Periodontal and Diabetes-Related Factors in the Diabetes and Periodontal Therapy Trial, A Randomized Controlled Trial. J Periodontol. 2016 Aug;87(8):900-13. doi: 10.1902/jop.2016.150727. Epub 2016 Apr 25. PMID 27108476
- [Derived] DPTT study group; Engebretson S, Gelato M, Hyman L, Michalowicz BS, Schoenfeld E. Design features of the Diabetes and Periodontal Therapy Trial (DPTT): a multicenter randomized single-masked clinical trial testing the effect of nonsurgical periodontal therapy on glycosylated hemoglobin (HbA1c) levels in subjects with type 2 diabetes and chronic periodontitis. Contemp Clin Trials. 2013 Nov;36(2):515-26. doi: 10.1016/j.cct.2013.09.010. Epub 2013 Sep 27. PMID 24080100